CLINICAL TRIAL: NCT03101319
Title: Role of Vitamin D Supplementation in First Episode Schizophrenia: A Double Blind Controlled Study
Brief Title: Role of Vitamin D Supplementation in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Psychiatry, Ranchi, India (Other)
Collaborators: University of Pittsburgh (Other); Dr. Ram Manohar Lohia Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Varun S Mehta, Assistant Professor of Psychiatry, Central Institute of Psychiatry, Ranchi, India
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1D43TW009114 (NIH)
Record Dates: First submitted 2017-03-29; First posted 2017-04-05 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Cholecalciferol; Hydroquinones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antipsychotic and Vitamin D3 (Experimental): Subjects randomised to vitamin D3 arm will receive a tablet containing 60,000 IU vitamin D3 starting from the first day of visit and then be taken by mouth on fixed days every week amounting to a total duration of 08 weeks. The subjects will continue to receive antipsychotics as per the decision of the treating team
  Interventions: Drug: Vitamin D3 cholecalciferol
- Antipsychotic and B Complex (Placebo Comparator): Subjects randomised to the B Complex arm will receive a tablet of identical size, shape, colour and weight starting from the first day of visit and then be taken by mouth on fixed days every week amounting to a total duration of 08 weeks. The subjects will continue to receive antipsychotics as per the decision of the treating team
  Interventions: Drug: B Complex Oral Tablet

INTERVENTIONS:
Drug: Vitamin D3 cholecalciferol — As mentioned in the description of the study arm
  Arms: Antipsychotic and Vitamin D3
Drug: B Complex Oral Tablet — As mentioned in the description of the study arm
  Arms: Antipsychotic and B Complex

SUMMARY:
The treatment of schizophrenia is challenging as the existing medications improve only the positive symptoms with the limited benefit on cognitive and negative symptoms which have a large bearing on the functional outcome. Recent research has suggested the association of low level of vitamin D with schizophrenia but studies are few and marred by mixed results. Thus, we propose to evaluate the effect of weekly vitamin D3 supplementation in patients with first-episode schizophrenia through a randomised doubled blind placebo controlled design.Fifty-six participants of either sex (19 - 50 years) with schizophrenia having vitamin D insufficiency/deficiency (< 30 ng/ml) will be randomly supplemented with Vitamin D3 or placebo for 8 weeks in 1:1 pattern. The clinical treatment i.e., antipsychotic medications will be continued as usual within the two groups. Participants in both the groups will be assessed at study entry, at the end of the 04 and 08 weeks (after completing supplementation) on the Positive and Negative Syndrome Scale (PANSS), Computerized Neurocognitive Battery (CNB) & Clinical Global Improvement (CGI) subscale (CGI-I). Raters will be blind to the group assigned to participants. Side effects will be monitored at every visit. The serum levels of vitamin D will be measured at baseline and at the end of 08 weeks.

DETAILED DESCRIPTION:
Patients diagnosed with schizophrenia as their first episode (<7 years' duration of illness) and receiving treatment from the Central Institute of Psychiatry, Ranchi will be invited for the study. The patients will be explained about the study and the patients giving the consent for the study will be screened for vitamin D3 insufficiency/deficiency. The patient would be selected for the study if 25 (OH) D is below 30 ng/ml and fulfils the clinical inclusion criteria. The patient would be recalled for enrolment in the study and the socio-demographic details will be collected along with the baseline evaluation. The patients will be randomized to either vitamin D3 or B-Complex group in a 1:1 proportion. Both the groups would be matched for age and gender as these may affect clinical outcome of schizophrenia and will balance the unknown confounding factors. The randomization scheme will utilize computer-generated random numbers that will be available with the PI who will supervise the dispensing the medication, the research assistant will be blind to the randomization numbers. This scheme will be stored in a password-protected computer and password-protected file. Only PI will have access to this file. The file will be opened only if a participant reports serious side effects. The double-blind design will be continued through the study period. The medications will be stored at room temperature and the investigators will supervise the dispensing of the study medication to subjects and/or their caregivers. Patients randomized to vitamin D3 arm will receive 4 tablets (containing 60,000 IU vitamin D3) on the first day of visit and after the fourth week (visit 3) respectively to be taken by mouth on fixed days every week. This dose is the recommended regimen by International Endrocrinological Society. The subjects will receive either vitamin D3 or B Complex weekly for 08 weeks along with the antipsychotic medications as determined by the treating team. The treating team will be encouraged to maintain stable doses if feasible. After the duration of 08 weeks, the dosage of vitamin D3 will be continued as per the serum levels and the recommendation guidelines whereas the antipsychotic medications will be continued as per the clinical response and decision of the treating team.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Either sex between 19-50 years
3. First episode schizophrenia with illness (< 7 years) receiving inpatient treatment
4. Serum (25) OH D below 30 ng/ml

Exclusion Criteria:

1. Presence of co-morbid psychiatric disorder
2. History of substance use meeting dependence criteria excluding caffeine
3. Co-morbid medical illness or medications known to affect vitamin D e.g. Hypothyroidism, Arthritis, Osteoporosis, Rickets, End Stage Renal Disease, Malabsorption Syndromes, Corticosteroid therapy
4. Patients already on Vitamin D supplementation
5. Patients with BMI more than 30kg/m² & women who have reached menopause as they have higher dietary requirements

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-05-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Change in the symptom dimensions of schizophrenia | Both the assessments (PANSS & CNB) would be done at baseline (at study entry) and repeated at the end of 4 weeks and 8 weeks respectively after receiving the study medication.
  The outcome would be assessed as a change in the positive symptoms, negative symptoms and cognitive symptoms of schizophrenia. The Positive and Negative Syndrome Scale (PANSS) would be used to evaluate the change in the positive symptoms and the negative symptoms. The Computerized Neurocognitive Battery (CNB) would be used to assess the change in the cognitive symptoms of schizophrenia

SECONDARY OUTCOMES:
Clinical Improvement | The assessment would be done at the end of 4 weeks and 8 weeks respectively after receiving the study medication.
  Clinical Global Impression - Improvement (CGI - I) sub domain of the scale will be used to assess the patient's global functioning after initiating the study medication.

OTHER OUTCOMES:
Side effects | Both the assessments would be done at baseline (at study entry) and repeated at the end of 4 weeks and 8 weeks respectively after receiving the study medication.
  The Vitamin D side effect check list will be administered to assess the adverse effects associated with vitamin D supplementation. The Liverpool University Neuroleptic Side Effect Rating Scale (LUNSERS) will be used to measure the severity of the neuroleptic side effects
Blood levels of serum 25 (OH) D, calcium & phosphorous | The blood would be drawn for assessment at the end of 8 weeks after receiving the study medications
  Blood sample will be collected early in the morning before breakfast by venipunture in a vacutainer (approx. 05 ml) for the assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Varun S Mehta, MD, Principal Investigator — Central Institute of Psychiatry; D Ram, MD, Study Chair — Central Institute of Psychiatry; Smita Deshpande, MD, Study Chair — Dr. Ram Manohar Lohia Hospital, and Post Graduate Institute of Medical Education and Research; Triptish Bhatia, PhD, Study Chair — Dr. Ram Manohar Lohia Hospital, and Post Graduate Institute of Medical Education and Research; Vishwajit L Nimgaonkar, MD, Study Chair — University of Pittsburgh
Locations (1):
- Central Institute of Psychiatry, Ranchi, Jharkhand, India

IPD SHARING:
Plan to Share IPD: No